CLINICAL TRIAL: NCT03610347
Title: Study to Evaluate the Efficacy and Safety of Paclitaxel Eluting Balloon After Bare Metal Stent Implantation Versus Drug-eluting Stent in St Elevation Myocardial Infarction
Brief Title: Paclitaxel Eluting Balloon After Bare Metal Stent Implantation vs. Drug-Eluting Stent in St Elevation Myocardial Infarction
Acronym: PEBSI-2
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low recruitment
Sponsor: Fundacion Investigacion Interhospitalaria Cardiovascular (Other)
Collaborators: Effice Servicios Para la Investigacion S.L. (Industry)
Responsible Party: Principal Investigator, Arturo García-Touchard, Principal Investigator, Fundacion Investigacion Interhospitalaria Cardiovascular
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PEBSI-2
Record Dates: First submitted 2018-07-26; First posted 2018-08-01 (Actual); Last update posted 2020-05-26 (Actual); Status verified 2020-05

CONDITIONS: Acute Myocardial Infarction
MeSH Terms: interventions — Drug-Eluting Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bare metal Stent plus Paclitaxel Balloon (Experimental): Conventional bare metal Stent plus Paclitaxel Eluting Balloon(Pantera Lux®)
  Interventions: Device: Bare metal Stent plus Paclitaxel Balloon
- Drug-Eluting Stent (DES) (Active Comparator): Sirolimus Eluting Stent (Orsiro®)
  Interventions: Device: Drug Eluting Stent

INTERVENTIONS:
Device: Bare metal Stent plus Paclitaxel Balloon
  Arms: Bare metal Stent plus Paclitaxel Balloon
Device: Drug Eluting Stent
  Arms: Drug-Eluting Stent (DES)

SUMMARY:
Study objective is the evaluation of safety and efficacy at 12 months of the combination treatment of bare metal Stent plus Paclitaxel Eluting Balloon vs drug eluting stent in patients with ST-elevation myocardial infarction with less than 12 hours of evolution.

DETAILED DESCRIPTION:
This is a multicenter, prospective, randomized, open study

After the permeabilization of the clinical event responsible artery patients will be randomized in a 1:1 ratio to one of the following treatment groups:

Group 1: insertion of a bare metal stent with post-dilatation with a paclitaxel eluting balloon (Pantera Lux ®)

Group 2: insertion of a drug elution stent

Patients (or their legal representative) must sign the consent before randomization.

Patients will be monitored 30 days after surgery, at 6 and 12 months.

The primary efficacy endpoint is Target Vessel Failure (TVF) at 12 months

This study will involve patients over 18 years old with STEMI, or new left bundle branch block or posterior AMI (ECG) that occur within 12 hours of onset of symptoms.

A total of 516 patients will be included.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged equal or older than 18 years.
* Acute myocardial infarction (AMI) within 12 hours of evolution (from the onset of symptoms) systolic time elevation of at least 1 mm (recorded in two or more contiguous leads), new left bundle branch block, or true posterior infarction.
* Patients candidates for primary angioplasty as medical criteria
* Written informed consent according to International Conference on Harmonization / Guide Clinical Practice and local legislation, obtained before any study procedure.
* Diameter vascular coronary artery to treat between 2 mm and 4 mm.
* Patients with 85-100% stenosis and TIMI Score (Thrombolysis In Myocardial Infarction) of 0-I.

Exclusion Criteria:

* Patients who refuse to participate in the study
* Cardiogenic shock (defined as systolic blood pressure less than 80 mm Hg for more than 30 minutes or need for vasopressors or intra-aortic balloon counterpulsation)
* Concomitant diseases associated with a life expectancy of less than one year
* Angiographic variables:

  * Trunk unprotected
  * Branching (side branch greater than 2.5 mm)
  * Sinus tachycardia segment elevation myocardial infarction thrombosis secondary to stent
  * If more than one stent to treat a single segment (overlapping stents)
  * Patient candidate for surgical revascularization within 30 days
  * Stenosis of greater than 30 mm in length (corresponding with the ball longer available)
  * More severe stenosis in the same artery in which is expected to be addressed in the next 9 months
* Women at childbearing age, where there is the possibility of pregnancy during the first year of follow-up, or nursing.
* Any clinical condition, which in the opinion of the investigator, is considered clinically significant as to participate in the study.
* Subjects who are participating in any study drug or medical.
* Individuals who show inability to follow instructions or help during the course of the study.
* Bleeding diathesis or other disorders such as gastrointestinal ulceration or cerebral circulatory disorders, restricting the use of treatments platelet aggregation inhibitors and anticoagulants.
* Patients with an ejection fraction <30% (if known).
* Allergy or hypersensitivity to paclitaxel intolerance, or compounds structurally related to the Butyryl tri-n-hexyl citrate (BTHC) matrix of administration.
* Severe allergy to contrast media.
* Coronary artery spasm in the absence of significant stenosis.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2016-06-29 (Actual); Primary Completion 2020-01-28 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Target Vessel Failure (TVF) | 1 year
  Efficacy: TVF define as a the composite of cardiac death, target-vessel myocardial infarction, or ischemia-driven target-lesion revascularization

SECONDARY OUTCOMES:
Target Lesion Revascularization (TLR) | 1 year
  Efficacy: ischemia-driven target-lesion revascularization
Major Adverse Cardiac Events (MACE) | 1 year
  Safety: Major Adverse Cardiac Events (MACE) at 12 months (death, re-infarction, acute cardiovascular disease, hemorrhagy and/or stent thrombosis).

OTHER OUTCOMES:
Angiographic Substudy | 9 months
  QCA late loss
Optical Coherence Tomography (OCT) Substudy | 3 and 6 months
  Stent struts coverage by intravascular OCT

CONTACTS AND LOCATIONS:
Locations (16):
- Spain (16):
  - H. U. Son Espases, Palma de Mallorca, Balearic Islands
  - H. U. Puerto Real, Puerto Real, Cádiz
  - H. U. de Bellvitge, L'Hospitalet de Llobregat, H. U. de Bellvitge
  - Complejo Hospitalario U. de Albacete, Albacete
  - H. del Mar, Barcelona
  - H. U. Vall D'Hebron, Barcelona
  - H. Clínic, Barcelona
  - H. General U. de Ciudad Real, Ciudad Real
  - H. U. Virgen de las Nieves, Granada
  - H. U. de La Princesa, Madrid
  - H. Clínico San Carlos, Madrid
  - H. U. 12 de Octubre, Madrid
  - H. U. Puerta de Hierro Majadahonda, Madrid
  - H. Regional U. de Málaga, Málaga
  - H. U. i Politècnic La Fe de Valencia, Valencia
  - H. Clínico U. de Valladolid, Valladolid

REFERENCES:
- [Derived] Garcia-Touchard A, Gonzalo N, Goicolea J, Gomez-Lara J, Martin-Yuste V, Peral V, Martinez-Romero P, Vaquerizo B, Sanchez-Recalde A, Sarnago F, Oteo JF, Alfonso F. Early coronary healing in ST segment elevation myocardial infarction: sirolimus-eluting stents vs. drug-coated balloons after bare-metal stents. The PEBSI-2 optical coherence tomography randomized study. Coron Artery Dis. 2021 Dec 1;32(8):673-680. doi: 10.1097/MCA.0000000000001038. PMID 33826537